CLINICAL TRIAL: NCT05696093
Title: Efficacy of Cotrimoxazole as a De-escalation Treatment of Ventilator-Associated Pneumonia in Intensive Care Unit. Multicentric Non-inferiority Randomised Controlled Trial
Brief Title: Efficacy of Cotrimoxazole as a De-escalation Treatment of Ventilator-Associated Pneumonia in Intensive Care Unit
Acronym: COTRIVAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220799
Record Dates: First submitted 2022-11-21; First posted 2023-01-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Associated Pneumonia
Keywords: intensive care unit; de-escalation; cotrimoxazole; Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Multicentre randomized non-inferiority trial comparing cotrimoxazole to standard antibiotic therapy for enterobacterial VAP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cotrimoxazole (Experimental): Use of cotrimoxazole for enterobacterial VAP. Posology and modalities of antibiotic administration will be optimized based on most recent recommendations for ICU patient. They will receive the treatment for 28 days or until death or until ICU discharge if its before 28days.
  Interventions: Drug: cotrimoxazole
- standard antibiotic therapy (Active Comparator): Use of standard antibiotic therapy enterobacterial VAP. Posology and modalities of antibiotic administration will be optimized based on most recent recommendations for ICU patient. They will receive the treatment for 28 days or until death or until ICU discharge if its before 28days.
  Interventions: Drug: standard antibiotic therapy

INTERVENTIONS:
Drug: cotrimoxazole — Use of cotrimoxazole therapy for enterobacterial VAP
  Arms: cotrimoxazole
Drug: standard antibiotic therapy — Use of standard antibiotic therapy for enterobacterial VAP
  Arms: standard antibiotic therapy

SUMMARY:
Efficacy of cotrimoxazole as a de-escalation treatment for adult patients Ventilator-Associated Pneumonia in intensive care unit Multicentre randomized non-inferiority trial comparing cotrimoxazole to standard antibiotic therapy for enterobacterial VAP

DETAILED DESCRIPTION:
Multicentre randomized non-inferiority trial comparing cotrimoxazole to standard antibiotic therapy for enterobacterial VAP. Selection of patients will be done by physicians in ICU. All clinically suspected VAP will be confirmed with a lung sample (preferably bronchoalveolar lavage or protected distal specimen, otherwise endotracheal aspiration). Patients with a microbiologically confirmed VAP due to an Enterobacteriaceae susceptible to cotrimoxazole and at least one antibiotic of the empiric antibiotic therapy (based on international recommendations) will be included. After written informed consent, they will be randomized (1:1), using a computer-generated randomization scheme of various-sized blocks, stratified by presence of septic shock at VAP diagnosis and by presence of COVID-19 pneumonia on ICU admission, through a centralized 24 hours internet service (CleanWEB™) to cotrimoxazole, or best standard of care (either a beta-lactam or a fluoroquinolone), after randomization for a total duration of 7 days (including empiric initial appropriate treatment). Posology and modalities of antibiotic administration will be optimized based on most recent recommendations for ICU patients. Because antibiotic therapy will be variable in the control group, single or double blind is not appropriate. Daily follow-up until death or ICU discharge or day 28 will be performed (vital status, antibiotic therapy, new infection, Clostridium-difficile infection). Clinical (arterial blood gas, temperature, haematology, tracheal secretions) and radiological cure (chest X-ray) will be assessed at Day 7. Systematic MDR bacteria screening will be performed weekly and at ICU discharge. Vital status will be assessed at day 90. Alive patients leaving ICU before 90 days will be contacted by phone (if discharge at home) or by interview at hospital (if transferred in a different ward). Assessment of the clinical and radiological cure by an independent committee (1 specialist in infectious disease and 1 intensivist), blinded of the randomization arm (PROBE methodology).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in an ICU
* Under mechanical ventilation for at least five days
* Microbiologically confirmed VAP preferably on a distal lung sample (bronchoalveolar lavage or protected distal specimen) otherwise endotracheal aspiration
* Enterobacteriaceae susceptible to cotrimoxazole, and for polymicrobial VAP, all bacteria susceptible to cotrimoxazole
* 5) Treated for at least 24 hours by an appropriate empiric antibiotic therapy (at least one effective antibiotic from the initiation of treatment for this VAP episode), and for polymicrobial VAP, all bacteria susceptible to empiric antibiotic therapy
* Stability of haemodynamic (stability or decrease in catecholamine dose) and respiratory (stability or improvement of FIO2) parameters

Exclusion Criteria:

* Haemodynamic instability (increasing dose of a catecholamine in the last 24 hours)
* Contra-indication to cotrimoxazole:

  * allergy,
  * advanced liver insufficiency,
  * renal dysfunction with clearance <15 mL/min/1.73 m² without hemodialysis
  * G6PD deficiency
  * history of hypersensitivity to one of the components (in particular, hypersensitivity to sulphonamides
  * known macrocytic anemia defined by VGM >
  * treatment with methotrexate
* Infection requiring prolonged antibiotic-therapy (pleural empyema, lung abscess, necrotizing pneumonia, etc…)
* Cystic fibrosis
* Immunosuppression (neutropenia, HIV with CD4 lymphocytes below 200/mm3, immunosuppressive therapy or corticosteroid therapy >0.5 mg/kg/j before ICU admission)
* Cardiac arrest without awakening
* Moribund state (patient likely to die within 24h)
* Limitation of life support (comfort care applied only) at the time of screening
* Enrolment to another interventional study on VAP care/management
* Pregnancy or breastfeeding
* Subject deprived of freedom, subject under a legal protective measure
* No affiliation to any health insurance system
* Refusal to participate to the study (patient or legal representative or family member or close relative if present)
* Patients previously included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that cotrimoxazole is non-inferior to best standard of care for the treatment of VAP in ICU in term of survival at day 28 | 28 days after inclusion
  Vital status at day 28

SECONDARY OUTCOMES:
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in term of mortality at day 90 | 90 days after inclusion
  Vital status at day 90
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in IC in terms of mechanical ventilation (MV)-free-days at day 28 | 28 days after inclusion
  number of MV-free-days through day 28
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of rate of cure between days 7 and 10 | days 7 and 10 after inclusion
  Clinical, biological and radiological cure evaluated 7 to 10 days after VAP diagnosis, defined as the combination of resolution of signs and symptoms present at enrolment, biological improvement, and improvement or lack of progression of radiological signs, as adjudicated by an independent committee (PROBE methodology)
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of VAP recurrence | 28 days after inclusion
  new episode of VAP with the same Enterobacteriaceae
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of ICU length of stay | 28 days after inclusion
  ICU length of stay
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of hospital length of stay | 28 days after inclusion
  hospital length of stay
To assess the safety of cotrimoxazole compared to best standard of care at day 28 in terms of allergy to antibiotics | 28 days after inclusion
  safety (rate of allergy due to antimicrobial drug)
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of mortality at day 28 | 28 days after inclusion
  Vital status at day 28
To demonstrate that cotrimoxazole is superior to best standard of care for the treatment of VAP in ICU in terms of overall antibiotic consumption | day 28 after inclusion
  antibiotic-free days at day 28
To assess the ecological impact of the treatment in terms of acquisition of MDR bacteria in ICU | 28 days after inclsuion
  evolution of rate of MDR bacterial colonization on systematic screening at enrolment until ICU discharge
To assess the ecological impact of the treatment in terms of rate of Clostridioides difficile infection | 28 days after inclusion
  diagnostic of Clostridioides difficile infection between inclusion and day 28

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - Médecine Intensive Réanimation - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Médecine Intensive Réanimation - Centre Hospitalier Universitaire Angers, Angers
  - Médecine Intensive Réanimation - Centre Hospitalier Béthune - Beuvry, Béthune
  - Réanimation Médico-chirurgicale - Hôpital Avicenne, Bobigny
  - Médecine Intensive Réanimation - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - Réanimation Médico-chirurgicale - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Réanimation polyvalente et Unité de surveillance continue - Centre Hospitalier de Cholet, Cholet
  - Réanimation Médicale - Centre Jean Perrin - Site Gabriel Montpied, Clermont-Ferrand
  - Médecine Intensive Réanimation - Hôpital Louis Mourier, Colombes
  - Réanimation polyvalente et surveillance continus - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Médecine Intensive Réanimation - Hôpital François Mitterrand, Dijon
  - Réanimation Polyvalente - Centre Hospitalier Annecy Genevois, Épagny
  - Médecine Intensive Réanimation - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Médecine Intensive Réanimation - Hôpital Michallon, La Tronche
  - Réanimation Médicale - Hôpital Robert Salengro, Lille
  - Réanimation médicale - Centre Hospitalier de Longjumeau, Longjumeau
  - Réanimation et Surveillance continue - Centre Hospitalier de Melun, Melun
  - Médecine Intensive Réanimation - CHRU de Nancy - Hôpitaux de Brabois, Nancy
  - Réanimation Médicale et Maladies Infectieuses - Hôpital Laennec, Nantes
  - Médecine Intensive et Réanimation - Hôpital de la Pitié Salpêtrière, Paris
  - Réanimation Médicale - Hôpital de la Pitié Salpêtrière, Paris
  - Réanimation Médicale - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Intercommunal Saint-Germain-en-Laye, Poissy
  - Médecine Intensive Réanimation - Hôpital René Dubos, Pontoise
  - Médecine Intensive Réanimation - Centre Hospitalier Léon Binet, Provins
  - Médecin Intensive Réanimation - Hôpital Delafontaine, Saint-Denis
  - Réanimation Polyvalente - Centre Hospitalier Universitaire Nord Saint-Etienne, Saint-Priest-en-Jarez
  - Médecine Intensive Réanimation - Nouvel Hôpital Civil, Strasbourg
  - Réanimation Polyvalente - Hôpital Sainte Musse, Toulon
  - Médecine Intensive Réanimation - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No